CLINICAL TRIAL: NCT03924258
Title: Study of the Prevalence of Iron Deficiency in Patients With Heart Failure
Acronym: CARENFER IC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: VIFORFRANCE (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CARENFER IC
Record Dates: First submitted 2019-04-18; First posted 2019-04-23 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HEART FAILURE (Experimental): Patients with Heart Failure diagnosis
  Interventions: Diagnostic Test: Iron status testing

INTERVENTIONS:
Diagnostic Test: Iron status testing — Blood sample for iron status testing

SUMMARY:
Despite its known prevalence in Heart Failure, a recent study conducted by Prof. Cacoub (unpublished) on the French national health insurance database showed that iron deficiency was a poorly diagnosed and poorly treated comorbidity. In chronic diseases including Heart Failure, Transferrin Saturation Factor is only performed in about 10% of cases while it is recommended for patients with Heart Failure (French Health High Authority 2011). The purpose of this study is to obtain current data on the prevalence of iron deficiency in France in patients with Heart Failure, applying the recommendations of European Society of Cardiology and French Health High Authority (determination of ferritinemia and Transferrin Saturation Factor).

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, over 18 years of age
* Patient present at the hospital on the day of the study
* Diagnosis of Heart Failure (acute or chronic) regardless of left ventricular ejection fraction (LVEF)
* Patient with signed consent

Exclusion Criteria:

* Protected patient: major under guardianship, tutorship or other legal protection, deprived of liberty by judicial or administrative decision
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1300 (Estimated)
Dates: Start 2019-05-15 (Estimated); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Complete blood iron status | One day
  ferritin, Transferrin Saturation Factor

IPD SHARING:
Plan to Share IPD: No